CLINICAL TRIAL: NCT05197816
Title: MotIoN aDaptive Deep Brain Stimulation for MSA
Acronym: MINDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Oxford University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20/LO/1034
Record Dates: First submitted 2021-11-29; First posted 2022-01-20 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-08

CONDITIONS: MSA - Multiple System Atrophy
Keywords: deep brain stimulation; autonomic
MeSH Terms: conditions — Shy-Drager Syndrome | interventions — Deep Brain Stimulation

STUDY DESIGN:
Intervention Model Description: Evaluation of symptomatology "on" and "off" adaptive deep brain stimulation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Deep brain stimulation (Experimental): All patients will undergo adaptive deep brain stimulation with results compared before and after stimulation
  Interventions: Device: Deep brain stimulation

INTERVENTIONS:
Device: Deep brain stimulation — Electrical pulses from implanted generator that adapts to patient activity and/or physiology

SUMMARY:
Patients routinely undergo deep brain stimulation (DBS) for treatment of symptoms related to neurodegenerative conditions, most commonly Parkinson's disease. In the Investigator's experience, and published evidence shows, that stimulation has effects on the autonomic nervous system. In patients undergoing therapeutic DBS for a particular subtype of Parkinsonism (Multiple System Atrophy), the effects on autonomic parameters such as blood pressure and bladder symptoms has been shown to be improved by the investigators (unpublished data). In this current study, the investigators plan to use a novel technique of adaptive DBS in order to provide stimulation dependent on patient physiological or positional factors. This is with the aim of making stimulation more responsive and patient-specific.

DETAILED DESCRIPTION:
Aim and patient group:

Multiple System Atrophy is a form of Parkinsonism and is a neurodegenerative condition that is characterized by gait and autonomic failure. The aim of this study is to assess the effects of aDBS of the Pedunculopontine Nucleus (PPN) on autonomic and gait symptoms in a group of 5 patients with MSA. Patients will enter our routine selection process but patients in the study will be selected for predominantly autonomic symptoms as per the inclusion criteria below. The aim is to test whether or not PPN aDBS improves quality of life, and has an effect on a variety of measurable autonomic parameters in this subset of patients. Secondary aims are to assess the safety of DBS in MSA, and to look at the structural projections and effects on brain networks associated with stimulation.

Background:

Deep Brain Stimulation (DBS) is a routine treatment for movement disorders such as Parkinson's disease (PD). In Oxford, around 80 DBS operations per year are performed, and approximately two thirds of these are in patients with PD. Multiple System Atrophy (MSA) is a 'Parkinsonian' condition similar to PD and is a progressive, incurable, neurodegenerative condition characterized by a combination of Parkinsonism, ataxia, and autonomic failure. Any one of these three features may predominate, making diagnosis difficult; however, virtually all patients have autonomic dysfunction. Indeed, autonomic dysfunction is the presenting feature in half of patients that have Parkinsonism or ataxia predominant MSA. The motor manifestations such as gait problems, ataxia, and postural abnormalities are very similar to those encountered by patients with Parkinson's disease, though unfortunately are usually less responsive to dopamine agonists and so can be more disabling. Patients tend to progress more quickly, often confined to a wheelchair within 3-5 years of diagnosis, and death is usually within a decade.

Whilst DBS has sometimes been performed for the treatment of MSA, including in Oxford , the primary outcome measure is usually the motor outcome, despite the fact that the autonomic symptoms are probably the predominant factor in causing a reduced quality of life. This is because DBS is traditionally used to control motor symptoms and the exploration of its effects on autonomic function are relatively new, and pioneered by the investigators.

The most common complaints caused by autonomic dysfunction in MSA are related to orthostatic hypotension and neurogenic bladder. The former causes dizziness, fatigue and, when a severe fall in BP occurs on standing, can lead to collapse. This may be, at least in part, a cause for the numerous falls that these patients suffer. Part of the aim of this study is to look at orthostatic BP changes with and without stimulation and see whether these are improved by DBS. This may correlate with a reduction in falls, although this study is unlikely to be powered to answer this specific question. Other 'autonomic' problems include bladder dysfunction, sleep disorders, exercise intolerance and problems with thermoregulation and sweating. These will be captured using questionnaires.

Regarding the target used for DBS, a well-established target to improve gait and postural abnormalities in PD is the pedunculopontine nucleus (PPN). It has been demonstrated that the PPN is also a brain area that, when stimulated, improves bladder function in these patients. It has also been shown that PPN stimulation reduces postural fall in BP in a group of PD patients treated primarily for gait and postural problems. Whilst these studies provide a rationale for looking at similar parameters in MSA patients, this study aims to answer the question as to whether it will work for these symptoms in MSA, in addition to the motor symptoms routinely treated.

The investigators have already shown in 5 patients with MSA that these symptoms are improved with PPN DBS. The difference in this trial is the usage of a new DBS device. This is a novel device where stimulation parameters can be changed in response to changes in the patient's position, activity, or physiological parameters.

Usage of adaptive stimulation:

The investigators intend to study the usage of motion-based control of stimulation. In the current trial, the main aim is to assess the effects of DBS on gait, sleep, and blood pressure control.

In previous studies, the investigators have noted that while standing, blood pressure is increased with stimulation, as is lying blood pressure. Supine hypertension may increase the stroke risk for these patients. Furthermore, the best improvement in gait is seen with a slightly different stimulation waveform.

In order to correct for this, the investigators propose to introduce motion-based adaptive stimulation which would involve the use of an accelerometer in changing between different stimulation parameters depending on the patient's position - so delivering a different waveform for lying and standing.

Justification/importance:

A trial of DBS to assess the effect on autonomic symptomatology of MSA has never been performed. We aim to combine a five patient clinical pilot study of DBS for MSA with an investigation of the neural circuitry underpinning autonomic control.

This translational strategy is likely to lead to a larger efficacy study of DBS for MSA as well as revolutionizing neural-based treatments in other autonomic disorders such as orthostatic hypotension and pure autonomic failure.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MSA with disabling autonomic symptoms
* >6/12 in the autonomic subsection (Q9-12) of the UMSAR scale
* Patient willing and able to give informed consent to involvement in the study.
* Male or female aged 55 years or over
* Able to walk (to perform gait analysis)
* Have an anticipated prognosis > 2 years

Exclusion Criteria:

* Female of child-bearing age
* The patient is unwilling to participate or unable to give informed consent.
* The patient has been deemed unfit for stimulator insertion by their healthcare team i.e. surgical contraindications to DBS:
* Bleeding or coagulation disorder
* Not fit for general anaesthetic
* Unable to deal with implanted DBS system (turn on and off and recharging where applicable, although it is acceptable if a carer can do this)
* Untreated anxiety or depression
* Unable to undergo preoperative MRI (e.g. metal implants)
* Subject is currently participating in a clinical investigation that includes an active treatment arm.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-12-03 (Actual); Primary Completion 2025-03-04 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Change in quality of life before and after DBS measured by EuroQol-5 domains | Pre-operative and at 3 months after stimulation
  EQ-5D before and after DBS. Each domain score 1-5, higher is worse.
Change in freezing of gait before and after DBS, measured by freezing of gait questionnaire | Pre-operative and at 3 months after stimulation
  Measured by Freezing of gait questionnaire (FOG) before and after DBS, Score 0-24, higher is worse.
Change in the number of sleep arousals per night | Pre-operative and at 3 months after stimulation
  Measured by change in number of arousals on polysomnography before and after DBS
Change in Cardiovascular symptoms following DBS (continuous blood pressure) | Pre-operative and at 3 months after stimulation
  24 hour ambulatory blood pressure recorded pre & 3 months post DBS
Change in Cardiovascular symptoms pre-post DBS (change in postural blood pressure) | Pre-operative and at 3 months after stimulation
  Measured by tilt table blood pressure, recorded pre & 3 months post DBS
Change of power in alpha bands on polysomnography before and after DBS | Pre-operative and at 3 months after stimulation
  Measured by change in alpha bands on polysomnography before and after DBS
Change of power in beta bands on polysomnography before and after DBS | Pre-operative and at 3 months after stimulation
  Measured by change in beta bands on polysomnography before and after DBS
Change of power in gamma bands on polysomnography before and after DBS | Pre-operative and at 3 months after stimulation
  Measured by change in gamma bands on polysomnography before and after DBS

SECONDARY OUTCOMES:
Number of patients with treatment-related adverse events | Throughout study up to 6 months
  Documentation of adverse events from intervention
Measurement of Falls frequency | Throughout study up to 3 months
  Falls diary
Frequency and volume of bladder voiding before and after stimulation | Pre-operative and at 3 months after stimulation
  British association of urological surgeons bladder diary
Autonomic function before and after stimulation measured by autonomic symptom profile | Pre-operative and at 3 months after stimulation
  Autonomic symptom profile questionnaire. Higher score is worse. Multiple sections, and composite score possible.
Carer Burden before and after stimulation measured by Zarit Burden interview | Pre-operative and at 3 months after stimulation
  Zarit Burden interview Carer Burden Questionnaire. Score 0-88, higher is worse.
MSA disease severity score before and after stimulation | Pre-operative and at 3 months after stimulation
  Unified MSA Rating Scale before and after stimulation. Scores 0-48 pt1, 0-56 pt2; higher is worse.
Gait Analysis before and after stimulation using gaitrite mat to measure gait and step velocity and symmetry | Pre-operative and at 3 months after stimulation
  Gait parameters testing using Gaitrite mat

CONTACTS AND LOCATIONS:
Locations (1):
- John Radcliffe Hospital, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Undecided We are recruiting only 5 patients, so sharing IPD even anonymised, may be identifiable. Decision will be taken when this can be definitively elucidated.